CLINICAL TRIAL: NCT03287479
Title: Prospective, Multi-center, Randomized, Controlled, Open Non-inferiority Trial Comparing a Semi-automated Closed Vitrification System (Gavi®) With a Manual Open Vitrification Sytem (Cryotop®)
Brief Title: Comparison of a Semi-automated Closed Vitrification System (Gavi®) With a Manual Open Vitrification Sytem (Cryotop®)
Acronym: Gavi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. M.Sc. Georg Griesinger, Prof. Dr. med. M.Sc., University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 712225
Record Dates: First submitted 2017-09-01; First posted 2017-09-19 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Infertility
Keywords: vitrification; semi-automated; manual
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Patients presenting ≥ 2 surplus regularly fertilized oocytes for cryoperservation on day 1 and patients undergoing elective cryopreservation of all available 2PN oocytes are are allocated to one of the two following procedures:
  Study group: surplus or all 2PN-stage oocytes are vitrified/warmed using the semiautomated Gavi® protocol.
  Control group: surplus or all 2PN-stage oocytes are vitrified/warmed using the manual Cryotop® protocol.
  Randomization will be performed on day of fertilization check by lab staff by opening a numbered, opaque sealed envelopes. The random sequence will be software-generated and blocks will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gavi® (Experimental): surplus or all fertilized oocytes will be cryoperserved by utilizing the closed, semi-automated Gavi® vitrification system
  Interventions: Procedure: Gavi® Vitrification
- Cryotop® (Active Comparator): surplus or all fertilized oocytes will be cryoperserved by utilizing the open, manual Cryotop® vitrification system
  Interventions: Procedure: Cryotop® Vitrification

INTERVENTIONS:
Procedure: Gavi® Vitrification — A closed, semi-automated vitrification system
  Arms: Gavi®
Procedure: Cryotop® Vitrification — An open, manual vitrification system
  Arms: Cryotop®

SUMMARY:
The GAVI® closed vitrification system is a CE labelled device licensed for use in human IVF. It has been developed to standardize the process of vitrification and to increase the safety of the procedure. It has been demonstrated that the novel semiautomated, closed vitrification system providing standardized equilibration prior to cryopreservation can produce similar results in terms of recovery rate and Embryo development up to the blastocyst stage as compared to the commonly used Manual Cryotop® open vitrifcation system when applied in a mouse model.

Furthermore, its application has resulted in first pregnancies after transfer of vitrifiedwarmed biopsied human blastocyts. Due to limitations of the preliminary studies (application in mouse model; absence of a larger clinical Trial assessing pregnancy and live birth rates in human model etc.) it is of paramount importance to compare the GAVI® vitrification method to the routinely used Cryotop® method in a human IVF setting employing randomization and a-priori sample size definitions.

The primary objective of this study is to demonstrate non-inferiority of vitrification using the semi-automated GAVI® closed system over the so-far routinely used manual Cryotop® open system in terms of post-thawing survival rate of 2PN oocytes.

The secondary objective of this trial is to study differences in embryo development, clinical pregnancy rate, ongoing pregnancy rate and live birth rate.

Furthermore, differences in procedure duration and convenience will be evaluated.

DETAILED DESCRIPTION:
One hundred and eighty (n=180) patients presenting more than 2 surplus 2 PNoocytes for vitrification or patients having all available 2PN oocytes electively vitrified will be randomly allocated (1:1) on day of fertilization check (day 1 after ovum pickup) to either procedure. In the study group, 2PN oocytes will be cryopreserved utilizing the semi-automated GAVI® open vitrification/warming technique.

In the control group, 2PN oocytes will be cryopreserved utilizing the manual Cryotop® open vitrification/warming technique.

The participation in this study will be limited to one cycle per patient. The study population consists of infertile couples undergoing IVF or ICSI treatment.

The study duration will be minimally 6 months per subject, e.g. the main study on the Primary outcome 2PN survival will be closed 6 months after randomization of the last patient.

Data from pregnancy and live birth outcome will be reported in addenda to the main clinical study report, as appropriate.

Before initiation of the study, all study sites will have investigators sufficiently trained.

The study will be performed in at least three sites within Germany. Patient recruitment will be competitive between study´centers.

The number of patients having oocyte pick-up during the time frame of the study conduct will consist of the population screened for inclusion.

In general, patients complying with the inclusion and exclusion criteria are eligible for inclusion and randomization.

There are no restrictions on the ovarian stimulation protocol and type or dose of ovulation induction agent (hCG or GnRH-agonist). Ovum pick-up is usually performed by transvaginal ultrasound-guided follicle aspiration 36±2 hours after hCG administration.

IVF or ICSI procedure is performed according to the investigator site´s standard operating procedure.

Fertilization check is performed on day 1 after ovum pick-up (OPU) 17±1 hours post insemination. The number of regularly fertilized oocytes, defined as oocyte presenting 2 pronuclei and 2 polar bodies, is assessed.

Patients presenting ≥ 2 surplus regularly fertilized oocytes for cryoperservation on day 1 and patients undergoing elective cryopreservation of all available 2 PN oocytes are are allocated to one of the two 2 procedures.

Randomization will be performed on day of fertilization check (day 1 after OPU) by lab staff by opening a numbered, opaque sealed envelopes. The random sequence will be software-generated and blocks will be used. All randomized patients will be logged in a paper- based randomization log with initials, DOB, study number, date, study group, name and signature of staff. Randomization will be stratified by Center and by indication (surplus 2PN oocyte cryopreservation vs. elective cryopreservation of all available 2PN oocytes).

All vitrification and warming procedures will be performed according to the manufacturer´s instructions.

In order to investigate the differences in vitrification procedure duration, the time span between starting with preparations needed for vitrification and transferring the vitrification device(s) into the liquid nitrogen tank for storage will be recorded.

Depending on the investigator site's cryo embryo transfer policy, in a subsequent natural or programmed cycle vitrified/warmed embryos will be replaced. Within site, all patients will undergo the same cryoprotocol for preparation of the endometrium.

There are no specifications on the protocol to be used. The number of 2 PN oocytes to be warmed will be decided by the investigator on a case by case basis. Embryo culture will be performed in all cases in individual microdroplets covered with culture oil up to the day of scheduled embryo transfer.

The day of embryo transfer and the number of embryos to be transferred will be decided by the investigator on a case by case basis.

In order to investigate survival rate, warmed 2PN-ooytes will be assessed immediately and 2 hours post warming procedure. Survival will be confirmed by the presence of an intact oolemma and regular cytoplasm 2 hours after the warming procedure and/or when embryonic cleavage is observed.

In order to investigate potential differences in development and quality of vitrified/warmed embryos cleavage and morphology will be assessed as followed:

day 2 (44±1 hours post insemination) : cell number, blastomere size, grade of fragmentation

day 3 (68±1 hours post insemination): cell number, blastomere size, grade of fragmentation

day 5 (116±1 hours post insemination): blastocyst stage (grade of expansion), ICM (inner cell mass) morphology, TE (trophectoderm) morphology

day 6 (140±1 hours post insemination): blastocyst stage (grade of expansion), ICM (inner cell mass) morphology, TE (trophectoderm) morphology

Patients who conceive will undergo ultrasound examination to confirm clinical pregnancy at 6-7 weeks of gestation. Follow-up data regarding the confirmation of ongoing pregnancy will be obtained by telephone. Live birth including related data will be obtained by a questonaire to be completed by the patient and returned to the investigator´s clinic.

The analyses will be done per-intention-to-treat (ITT) and per protocol (PP), as appropriate. The ITT population is the randomized patient population. The PP population is the population of patients undergoing an attempt of thawing.

Source data will be paper-based case report forms (CRF).

* study ID number
* date of birth (female patient)
* age female (years)
* age male (years)
* type of stimulation protocol (Antagonist/Agonist protocol, short/long protocol)
* type of gonadotropin used (uFSH, rFSH, HMG, mix, Elonva)
* total dose of gonadotropins
* type of oocyte insemination (IVF, ICSI)
* Date and time of trigger
* Type and dose of triggering medication
* Date and time of ovum pick-up
* Date of randomization
* study group
* date and time of IVF/ICSI
* date and time of fertilization check (2PN assessment)
* number of fertilized oocytes (2PN oocytes)
* reason for vitrification (surplus vs. elective)
* date and time of vitrification (start/end)
* duration of vitrification procedure (minutes)
* date and time of warming (start/end)
* duration of warming procedure (minutes)
* number of warmed 2PN-oocytes
* number of vital 2PN-oocytes
* number of top quality embryos on day 2, day 3, day 5 and day 6 (depending on day of embryo transfer)
* number of transferred embryos
* number of revitrified embryos
* cycle outcome (no pregnancy, positive hCG test)
* course of pregnancy (abortion, termination, vanishing twin, etc.)
* Multiplicity (singleton, twin, triplet)
* pregnancy outcome (clinical pregnancy, ongoing pregnancy, live birth)

Descriptive statistics will be performed by analysing median, mean, n, standard deviation, ranges and 95% confidence intervals (CI). The differences between arms will be summarized as absolute difference with 95% CI. For the primary outcome, a linear model will be constructed accounting for treatment group, study site and randomization stratum exclusively for the per-protocol population.

For secondary outcomes ITT and/or PP analyses will be performed. No correction for multiplicity is planned. Parametric and non-parametric tests will be used for normally distributed and non-normally distributed variables, respectively, to compare secondary outcomes between groups.

The patient data will be entered into a computer database in a pseudonymized way. Data management and analysis will be carried out by the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* IVF or ICSI treatment
* 2 or more surplus 2 PN oocytes OR elective cryopreservation of all 2 PN oocytes on day of fertilization check
* willingness to participate (signed ICF)

Exclusion Criteria:

* history of low response to controlled ovarian hyper stimulation in previous IVF or ICSI treatments (ESHRE Bologna criteria; Ferranetti et al., Hum Reprod 2011)
* uterine pathology evident on transvaginal sonography, hysterosalpingography, hysteroscopy or laparoscopy
* participation in a PGS or PGD program
* previous participation in this study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
post-thawing survival rate | 2 hours
  confirmation of survival by presence of intact oolemma and regular cytoplasm 2 hours post warming procedure and by observation of embryonic cleavage on

SECONDARY OUTCOMES:
Number of top quality embryos on day 2 | 2 days
  Number of top quality embryos on day 2 (according to the Istanbul Consensus on embryo assessment) divided by the number of vitrified- warmed 2PN-oocytes
Number of top quality embryos on day 3 | 3 days
  Number of top quality embryos on day 3 (according to the Istanbul Consensus on embryo assessment) divided by the number of vitrified- warmed 2PN-oocytes
Number of top quality embryos on day 5 | 5 days
  Number of top quality embryos on day 5 (according to the Istanbul Consensus on embryo assessment) divided by the number of vitrified- warmed 2PN-oocytes
Number of top quality embryos on day 6 | 6 days
  Number of top quality embryos on day 6 (according to the Istanbul Consensus on embryo assessment) divided by the number of vitrified- warmed 2PN-oocytes
Clinical pregnancy rate | 6 weeks
  number of viable pregnancies at 6 weeks of gestation per ITT and PP
Ongoing pregnancy rate | 12 weeks
  number of viable pregnancies at 12 weeks of gestation per ITT and PP
Live birth rate | 44 weeks
  number of at least one live born infant per ITT and PP

OTHER OUTCOMES:
Procedure duration | 1 day
  time span start - end of procedures in minutes:seconds, adjusted for number of 2 PN oocytes vitrified
Convenience | 1 day
  questionaire to be completed by operating lab personnel after having performed at least 3 procedures with both methods

CONTACTS AND LOCATIONS:
Overall Officials: Georg Griesinger, Prof Dr MSc, Principal Investigator — University of Luebeck
Locations (3):
- Germany (3):
  - Universitäres Kinderwunschzentrum Kiel, Kiel
  - Universitäres Kinderwunschzentrum Lübeck, Lübeck
  - Kinderwunsch-Zentrum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymized data can be shared after primary publication upon reasonable request.
Supporting Information: Study Protocol, CSR
Time Frame: from 12/2021 on
Access Criteria: https://bmcmedicine.biomedcentral.com/articles/10.1186/s12916-015-0532-z

REFERENCES:
- [Background] Roy TK, Brandi S, Tappe NM, Bradley CK, Vom E, Henderson C, Lewis C, Battista K, Hobbs B, Hobbs S, Syer J, Lanyon SR, Dopheide SM, Peura TT, McArthur SJ, Bowman MC, Stojanov T. Embryo vitrification using a novel semi-automated closed system yields in vitro outcomes equivalent to the manual Cryotop method. Hum Reprod. 2014 Nov;29(11):2431-8. doi: 10.1093/humrep/deu214. Epub 2014 Aug 27. PMID 25164022
- [Derived] Hajek J, Baron R, Sandi-Monroy N, Schansker S, Schoepper B, Depenbusch M, Schultze-Mosgau A, Neumann K, Gagsteiger F, von Otte S, Griesinger G. A randomised, multi-center, open trial comparing a semi-automated closed vitrification system with a manual open system in women undergoing IVF. Hum Reprod. 2021 Jul 19;36(8):2101-2110. doi: 10.1093/humrep/deab140. PMID 34131726
- See also: Hobson N, Filipovits J, Roy T, Brandi S, Woolcott R, Bowman M, McAthur S. First pregnancies from human embryos vitrified-warmed using the semi-automated GAVI® closed vitrification system. Hum Reprod 2016;31(1):i203-i204 — https://www.eshre.eu/Annual-Meeting/Helsinki-2016/Abstract-book.aspx